CLINICAL TRIAL: NCT05387356
Title: Evaluation of the Efficiency and Complications of the Consequtive Proning in Covid -19 ICU: A Retrospective Study
Brief Title: Evaluation of the Efficiency and Complications of the Consequtive Proning in Covid -19 ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, ESRA OZAYAR, Clinical Assoc. Prof , Anesthesiology and Reanimation Department, Kecioren Education and Training Hospital
Other Study IDs: Prone Position
Record Dates: First submitted 2022-05-23; First posted 2022-05-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19 Respiratory Infection
Keywords: prone position; intensive care unit
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prone position — thirty-one patients who had a positive test result for SARS-CoV-2 RNA through nasopharyngeal swab and underwent three subsequent prone positions for 16 hours will be enrolled the study. Medical datas of the patients will be obtained from patients' files which are strictly filled during pandemic. Prone position indication of intensive care unit (ICU) is in case of severe ARDS with PaO2/FiO2 <150 despite a PEEP >10 cmH2O.

SUMMARY:
Thirty -one confirmed Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2 ) infected patients with Acute Respiratory Distress Syndrome (ARDS) and placed in prone position(PP) for 3 times (PP1, PP2, PP3)consecutively will be included. Arterial blood gases (ABG), partial pressure of arterial oxygen/ fraction of inspired oxygen (PaO2/FiO2 ) ratios, partial pressure of carbondioxide (PaCO2), positive end expiratory pressure (PEEP), and fraction of inspired oxygen (FiO2) values will be recorded before (bPP), during (dPP)and after (aPP) every prone positioning. Eye, skin, nerve and tube complications related to prone positions wll be recorded

ELIGIBILITY:
Inclusion Criteria:

a positive test result for SARS-CoV-2 RNA through nasopharyngeal swab and underwent three subsequent prone positions for 16 hours will be enrolled the study. -

Exclusion Criteria:

negative test result for SARS-CoV-2 RNA -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Intensive care patient population who were intubated a positive test result for SARS-CoV-2 RNA through nasopharyngeal swab and underwent three subsequent prone positions for 16 hours will be enrolled the study. -
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
effects of prone position | 15 days
  The investigators will evaluate the arterial blood gase results and ventilator settings before after and during prone position

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No